CLINICAL TRIAL: NCT05573516
Title: A Comparative Study Between Positional and Lag Screws for the Fixation of Medial Malleolar Fractures
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kasr El Aini Hospital (Other)
Responsible Party: Principal Investigator, Ahmed Omar Sabry, Principal Investigator, Kasr El Aini Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AOS12345
Record Dates: First submitted 2022-10-05; First posted 2022-10-10 (Actual); Last update posted 2022-10-10 (Actual); Status verified 2022-10

CONDITIONS: Medial Malleolus Fracture; Ankle Fractures
MeSH Terms: conditions — Ankle Fractures | interventions — Open Fracture Reduction; Fracture Fixation, Internal

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fixation with 4mm lag screws (Experimental)
  Interventions: Procedure: Open reduction and internal fixation
- Fixation with 4mm fully-threaded positional screws (Active Comparator)
  Interventions: Procedure: Open reduction and internal fixation

INTERVENTIONS:
Procedure: Open reduction and internal fixation — unicortical fully threaded 4mm screws will be used as positional screws after completely reducing the fracture

SUMMARY:
A clinical trial comparing the outcomes of fixation of medial malleolar fractures either by fully threaded uni-cortical 4mm positional screws vs 4mm lag screws.

DETAILED DESCRIPTION:
Ankle fractures are one of the most common traumatic injuries an orthopedic surgeon encounters during their clinical practice, Hence looking into the best management of them and conducting extensive research to determine the best methods of their fixation would be justifiable. Malleolar fractures and in particular medial malleolar involve the articular surface of the ankle joint and hence a displacement beyond > 2mm requires careful anatomical restoration through open reduction and internal fixation. The medial malleolus is characterized with it's porous cancellous bone, and hence a lack of a secure fixation method is a major issue and is responsible for post-operative complication and delayed healing. The AO recommends fixation of these fractures with 4mm partially threaded lag screws. Some studies have arisen that may challenge this AO philosophy and raise the question if this actually is the best choice of treatment for medial malleolar fractures. The problem with lag screws is that they have a higher chance of unravelling. and other studies have shown that constructs fixated with fully threaded screws provide higher stability and provides higher shear resistanceand a higher pull-out strength. The other alternative to using a partially threaded lag screw would be a fully threaded lag screw of virtually the same length however it would act as a positional screw and hence the fracture displacement must be perfectly reduced with bone reduction forceps before inserting the fully threaded screws to achieve their property as positional screws.

A study conducted by parker et al. comparing the use of partially threaded and positional(fully threaded) screws of the same length found that compression force was in favor of the fully threaded screws. This could be due to threads of the fully threaded screws obtaining purchase in the dense physeal scar area while in the partially threaded screw, the threads bypass this physeal scar. Despite all this evidence and the widespread of this fracture among the population, the number of studies comparing lag vs positional screws in medial malleolar fractures is scarce and to our knowledge as of the time of the submission of this study, only a single study was made by Sayyed-Hosseinian et al., was performed as a pilot study comparing both fixation methods, due to the relatively small sample size , it indicates that further clinical trials are necessary to reach a reliable conclusion. The conduction of a clinical trial with a proper sample size should be done to assess if lag screws are actually a superior method to be considered the main recommendation, as the AO suggests, to treat medial malleolar fractures or if alternatively, positional screws are better, as some biomechanical tests mentioned prior have shown. This study will compare both methods to decide the superior fixation method in terms of achieving a better and faster quality of life post-surgery and and the least risk for potential complication for medial malleolar fractures by obtaining the AOFAS, MOXFQ and OMAS scores and comparing complications in both study groups.

ELIGIBILITY:
Inclusion Criteria:

•Displaced medial malleolar fractures (Herscovici type B and C) that can be fixed with screws.

Exclusion Criteria:

* Open fractures,
* Age <18 or > 70,
* Pathological fractures,
* Patients with DM,
* Type A and D fractures according to the Herscovici system(As these fractures would require screws to be positioned horizontally),
* associated tibial plafond fractures

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2022-08-18 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
AOFAS score | 6 wks (this time when the fracture has usually healed and the patients cat bear weight on the limb)

CONTACTS AND LOCATIONS:
Locations (1):
- Kasr Al Ainy-Cairo University- Faculty of Medicine, Cairo, Manial, Egypt

IPD SHARING:
Plan to Share IPD: Undecided